CLINICAL TRIAL: NCT00607802
Title: White Cell Transfer as Cancer Therapy
Brief Title: Donor White Blood Cell Infusion in Treating Patients With Metastatic or Unresectable Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CCCWFU-99107; CDR0000584624 (Registry Identifier: PDQ (Physician Data Query)); IRB00002178
Record Dates: First submitted 2008-01-30; First posted 2008-02-06 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Polymerase Chain Reaction

INTERVENTIONS:
Biological: leukocyte therapy
Genetic: polymerase chain reaction

SUMMARY:
RATIONALE: White blood cells from donors may be able to kill cancer cells in patients with cancer.

PURPOSE: This clinical trial is studying the side effects of donor white blood cell infusion in treating patients with metastatic or unresectable cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of white blood cell infusion in patients with metastatic or unresectable cancer.

Secondary

* Determine the efficacy of this therapy in these patients.

OUTLINE: Patients receive allogeneic white blood cell infusions once daily for 5-10 infusions.

Patients undergo blood sample collection periodically for correlative laboratory studies. The samples are evaluated by in vitro white cell kill assay before the first infusion, immediately after the first infusion, on day 2, and then immediately after the last infusion to assess in vitro cancer cell killing activity. Chimerism studies are performed before the first infusion, immediately after the first infusion, and then on days 2 and 7. Complete chimerism is assayed by short tandem repeat analysis using PCR. Patients with readily accessible tumor tissue (e.g., cervical or axillary lymph nodes or subcutaneous tumor nodules) may also undergo biopsy during the first week of treatment to demonstrate the presence or absence of tumor infiltrating granulocytes.

After completion of study therapy, patients are followed periodically for 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignancy

  * Metastatic or unresectable disease
  * Standard curative or palliative measures do not exist or are no longer effective
* Measurable or non-measurable disease

  * Measurable disease is defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
  * Non-measurable disease is defined as all other lesions (including small lesions and truly non-measurable lesions), including any of the following:

    * Bone lesions
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* No brain metastasis
* Healthy blood donor available meeting the following criteria:

  * Willing to be included in the White Cell Donor Registry created for this study
  * Willing to undergo granulocyte apheresis at the American Red Cross
  * ABO compatible with the patient
  * HLA-mismatched with the patient
  * Demonstrates ≥ 60% cytotoxic killing activity (CKA) as determined by in vitro white cell kill assay

    * Less than 60% CKA allowed if deemed suitable by the investigators

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 4 months
* ANC ≥ 1,000/µL
* Platelet count > 100,000/µL (platelet transfusion independent)
* Serum bilirubin ≤ 2 mg/dL
* AST and ALT < 3 times upper limit of normal
* Serum creatinine ≤ 2 mg/dL
* No uncontrolled diabetes mellitus
* No myocardial infarction within the past 30 days
* No active serious infection
* No HIV infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Negative panel reactive antibody test (i.e., absence of serum HLA antibody)

PRIOR CONCURRENT THERAPY:

* No prior fludarabine phosphate
* No prior stem cell transplantation
* At least 4 weeks since prior medical therapy, radiotherapy, or surgery
* More than 30 days since prior immunosuppressive agents other than steroids

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Response (complete response, partial response, stable disease, or disease progression)

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Cui, MD, PhD, Study Chair — Wake Forest University Health Sciences